CLINICAL TRIAL: NCT05163002
Title: Effectiveness of Nutrition Education in Carbohydrate Counting, in a Group Context, on Glycemic Control in People With Type 1 Diabetic
Brief Title: Effectiveness of Nutrition Education in Carbohydrate Counting in People With Type 1 Diabetic
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Universidade Nova de Lisboa (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Universidade Nova de Lisboa
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Experimental): Intervention arm, uncontrolled
  Interventions: Behavioral: Nutritional education & carbohydrate counting

INTERVENTIONS:
Behavioral: Nutritional education & carbohydrate counting — Nutrition Education with a multidisciplinary team

SUMMARY:
Carbohydrates are the nutrient in the diet with the greatest impact on blood glucose. Inadequate carbohydrate counts are associated with higher A1c and greater variations in postprandial blood glucose. Clinical guidelines for the nutritional treatment of diabetes recommend that patients with DM1 learn carbohydrate counting or some similar systematic strategy that allows for better metabolic control. However, despite the recommendations, this is still not a reality for most healthcare services treating individuals diagnosed with DM1.

DETAILED DESCRIPTION:
The study aims to assess the impact of a structured nutrition education programme for nutritional education and carbohydrate counting, in group sessions, on glycemic control and nutritional literacy in people with DM1. This will be achieved by evaluating the glycaemic control through A1c and daily glycaemic variability (time on target, mean glycaemia), as well as the level of knowledge before and after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged ≥18 years old who have been diagnosed with type 1 diabetes or parents of children and adolescents (< 18 years old) who have been diagnosed with type 1 diabetes;
* To be under intensive insulin therapy (basal/bolus system);
* To regularly use a continuous glucose monitoring system as primary method for glycaemic control;
* To be able to read and write.

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2023-04-30 (Estimated)

PRIMARY OUTCOMES:
Differences between baseline A1c (%) and 90 days after the last educational session. | 90 days
  The outcome will be assessed through blood exams

SECONDARY OUTCOMES:
Difference in the level of nutritional knowledge assessed through a questionnaire "Nutrition knowledge" collected at baseline and in the last educational session (scale 0 to 23, where 23 is the highest). | 90 days
  The level of knowledge will be measure in a likert scale from 0 (minimum) to 23 (maximum), where a higher score is better than a lower one
Difference in time in range (%) between baseline and 90 days following the last educational session | 90 days
  The outcome will be assessed through data from participants' continuous glucose monitoring system
Difference in the glucose coefficient of variation (%) between baseline and 90 days following the last educational session | 90 days
  The outcome will be assessed through data from participants' continuous glucose monitoring system
Difference in mean glycaemia (mg /dL) between baseline and 90 days following the last educational session | 90 days
  The outcome will be assessed through data from participants' continuous glucose monitoring system

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Medical School, Lisbon, Portugal